CLINICAL TRIAL: NCT02889458
Title: Preventing Breast Cancer in Hong Kong Chinese Women Through Personalized Risk Stratification and Characterization: an Epidemiologic Modeling Study and the Development of a Biorepository of Cases and Controls
Brief Title: Hong Kong Breast Cancer Study
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Gabriel Matthew Leung, Dean, Li Ka Shing Faculty of Medicine, The University of Hong Kong
Other Study IDs: BrCA.risk.001
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Ductal Carcinoma In Situ
Keywords: Chinese; Breast Cancer; Women
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood, normal breast tissue, and tumour tissue.

GROUPS / COHORTS (2):
- Case: Inclusion Criteria
  * Female
  * aged 18 or above
  * Chinese
  * Usually residing in Hong Kong (Definition: Having stayed in HK for at least three months during the six months before the reference time-point)
  * Able to speak Cantonese
  * Newly diagnosed with breast cancer or DCIS in 24 weeks
  Exclusion Criteria
  - Undergoing treatment for any non-breast cancer
  Subjects will complete a structured interview with a questionnaire with research assistants' aid. Specimen of blood, normal breast tissue and tumour tissue will be collected.
  Interventions: Other: Not Provided
- Control: Inclusion Criteria
  * Female
  * aged 18 or above
  * Chinese
  * Usually residing in Hong Kong
  * Able to speak Cantonese
  Exclusion Criteria
  - History of any cancer
  Subjects will complete a structured interview with a questionnaire with research assistants' aid. Specimen of blood will be collected.
  Interventions: Other: Not Provided

INTERVENTIONS:
Other: Not Provided

SUMMARY:
Introduction: With population ageing and increasing Westernization breast cancer continues to be important health conditions among women in Hong Kong. Greater collaborative research efforts are needed to examine the questions about population screening for breast cancer, the aetiology of such lesions and outcomes of breast cancer during survivorship period. There is a lack of locally-relevant models for assessing breast cancer risk. Contribution of novel genetic factors to breast cancer, identification of the key and functional alleles in gene regions associated with risk of breast cancer as well as gene-environment interaction, requires further investigation in Chinese population. Prognostic research studies in the West may not be readily applicable to the Chinese population.

Objectives: We aim to investigate the aetiology and outcomes of breast cancer in local Chinese by using case-control and cohort study design in the health care setting in Hong Kong. We aim to examine potential risk factors/biomarkers (both traditional and novel), and to build infrastructure and biobank for breast cancer surveillance. We will follow up cases prospectively as a survivor cohort.

Methods: A hospital-based case-control study and a prospective survivor cohort study will be conducted. Consecutive incident breast cancer and DCIS cases (n=3,501) within a 36-month period in Hong Kong were recruited from public hospitals, private hospitals and private practices; and controls were selected by frequency-matching on factors such as age and hospital/clinic setting, whenever possible. Cases will be prospectively followed up over a 10-year period, and data collection will occur at baseline (within 24 weeks of diagnosis), 3, 5 and 10 years following baseline assessment. Biologic samples (including both blood, and tumour and normal breast tissue samples from the cases, and blood samples from the controls) will be collected for later genetic and molecular study including WGS, GWAS, gene-environment interaction and molecular functional studies. Depending on availability of pathology samples and resources, additional studies such as tissue microarray block production will be considered and performed in future. Data will be analysed by traditional regression, EWAS and genetic association methods, whenever relevant.

Public Health Implications: The repository of clinical, radiological and biological materials assembled through this case-control study will serve as a common, publicly accessible platform for subsequent functional analysis and scientific interrogation. The case-control findings would offer an improved understanding to the state of the science on aetiology of breast cancer in Chinese women. In the genomics analysis, potential refined classification of breast tumours may enhance our understanding, detection and follow-up of such lesions, as well as enable us to have more informed targeted and personalized treatment selection for our women population. The cohort study findings are important for developing an effective strategy for the improvement of overall survival and quality of life for the cancer survivors in Chinese population.

ELIGIBILITY:
Case Inclusion Criteria:

* Female
* aged 18 or above
* Chinese
* Usually residing in Hong Kong (Definition: Having stayed in HK for at least three months during the six months before the reference time-point)
* Able to speak Cantonese
* Newly diagnosed with breast cancer or DCIS in 24 weeks

Case Exclusion Criteria:

* Undergoing treatment for any non-breast cancer

Control Inclusion Criteria

* Female
* aged 18 or above
* Chinese
* Usually residing in Hong Kong
* Able to speak Cantonese

Control Exclusion Criteria

- History of any cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese female who usually reside in Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
probability of developing breast cancer | 2 years
  We will estimate individualized breast cancer probabilities based on information on relative risks and the baseline hazard rate in Hong Kong Chinese women population. Risk factors will include age, age at menarche, age at first birth, family history of breast cancer, prior breast benign disease diagnosis, menopausal status, dietary pattern. Structured interviews will be provided by our trained interviewers to collect these data by using our survey questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel M Leung, MD, Principal Investigator — Li Ka Shing Faculty of Medicine, The University of Hong Kong
Locations (21):
- Hong Kong (21):
  - Baptist Hospital, Hong Kong
  - Caritas Medical Centre, Hong Kong
  - Evangel Hospital, Hong Kong
  - Grantham Hospital, Hong Kong
  - HK Sanatorium and Hospital, Hong Kong
  - Kwong Wah Hospital, Hong Kong
  - North District Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Pok Oi Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Ruttonjee Hospital, Hong Kong
  - St. Paul's Hospital, Hong Kong
  - St. Teresa's Hospital, Hong Kong
  - Tseng Kwan O Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Union Hospital, Hong Kong
  - United Christian Hospital, Hong Kong
  - Yan Chai Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol: BrCA.risk.001 — http://www.hkuctr.com/Study/Show/b122235f3995420a97d570a85d03b542